CLINICAL TRIAL: NCT02173834
Title: Activation of Brown Adipose Tissue in Lean and Obese Men
Brief Title: Brown Adipose Tissue and Body Mass Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, F Holleman, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL41577.018.12 METC 2012.214
Record Dates: First submitted 2014-03-20; First posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Obesity; Type 2 Diabetes Mellitus
Keywords: Brown Adipose Tissue; Weight; Sympathetic Nervous System
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lean subjects (Other): Lean, young, healthy, Caucasian, male subjects
  Interventions: Other: 18F- fluorodeoxyglucose-positron emission tomography Computed Tomography scan and 123I-metaiodobenzylguanidine-single-photon emission computed tomography scan
- Obese subjects (Other): Obese, Young, Healthy, Caucasian, male subjects
  Interventions: Other: 18F- fluorodeoxyglucose-positron emission tomography Computed Tomography scan and 123I-metaiodobenzylguanidine-single-photon emission computed tomography scan

INTERVENTIONS:
Other: 18F- fluorodeoxyglucose-positron emission tomography Computed Tomography scan and 123I-metaiodobenzylguanidine-single-photon emission computed tomography scan

SUMMARY:
In this study the investigators aim to investigate whether the sympathetic stimulation of BAT, as assessed with a 123I-metaiodobenzylguanidine single-photon emission computed tomography computed tomography scan, differs between lean and obese individuals, as an explanation for the diminished metabolic brown adipose tissue activity in obese subjects.

The investigators hypothesis is that sympathetic nervous system activity in the obese is diminished as compared to their leaner counterparts as an explanation for the diminished metabolic brown adipose tissue activity in the obese.

DETAILED DESCRIPTION:
The sympathetic nervous system is the primary activator of Brown Adipose Tissue.

Obese humans are known to have less metabolically active brown adipose tissue as compared to their leaner counterparts.

The reason for this diminished metabolic brown adipose tissue activity is unknown.

However, a lower sympathetic nervous system activation to brown adipose tissue in the obese might explain a diminished metabolic brown adipose tissue.

Therefore, in this study, both the sympathetic nervous system activation to brown adipose tissue and the metabolic activity will be measured in lean and obese subjects.

sympathetic nervous system activity will be measured using 123I-metaiodobenzylguanidine single-photon emission computed tomography scans, metabolic activity will be measured using 18F- fluorodeoxyglucose positron emission tomography CT scans.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Caucasian origin
* Subjects should be able and willing to give informed consent
* 18-40 years old
* BMI range of 19-25 kg/m2 (lean study subjects) or 28-40 kg/m2 (obese study subjects)

Exclusion Criteria:

* Renal failure (creatinine>135mmol/l)
* Daily use of prescription medication

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Difference in sympathetic stimulation to BAT between lean and obese individuals | Participants will be followed for a mean duration of 2 weeks (the maximal time period between the two scans) The outcome measurements will be assessed when the last subject has been scanned approximately one year after starting the trial

SECONDARY OUTCOMES:
Difference in correlation between sympathetic stimulation of BAT as assessed with 123I-MIBG SPECT scans and metabolic BAT activity as assessed with 18F-Fluorodeoxyglucose(FDG)- positron emission tomography(PET)-CT scan in lean and obese individuals | Participants will be followed for a mean duration of 2 weeks (the maximal time period between the two scans) The outcome measurements will be assessed when the last subject has been scanned approximately one year after starting the trial.
  The difference in correlation between sympathetic stimulation of BAT and metabolic BAT activity between lean and obese individuals.

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands